CLINICAL TRIAL: NCT06714188
Title: Application of Personalized Palliative Care in Patients With Newly Diagnosed Idiopathic Pulmonary Fibrosis - An Exploratory-Descriptive Study
Brief Title: Application of Personalized Palliative Care in Patients With Newly Diagnosed Idiopathic Pulmonary Fibrosis
Acronym: IPF-PPC
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: IPF-PPC
Record Dates: First submitted 2024-11-28; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-10

CONDITIONS: IPF
Keywords: Questionnaire; Palliative Care; IPF

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to develop a tool that helps the medical-nursing team in the identification of the real palliative care needs of each individual patient. Patients with newly diagnosed Idiopathic Pulmonary Fibrosis will be asked just a few simple questions in order to place them at the most appropriate level of palliative care (PC) even before the first medical contact. This would not only optimize resource allocation (e.g., allowing patients with low palliative needs to be assessed solely by the PC nurse), but also benefit patients who have difficulty leaving their homes by enabling them to receive evaluation and palliative care directly at home rather than after a hospital assessment.

DETAILED DESCRIPTION:
The population of this study consists of patients with newly diagnosed Idiopathic Pulmonary Fibrosis (IPF) who are being followed at the specialized outpatient clinics of APPI Fibrosi, within the Unit of Pulmonology and Respiratory Intensive Care, at the IRCCS Azienda Ospedaliero-Universitaria, Policlinico di S. Orsola.

During the initial interview prior to the pulmonology visit, Pulmonologist A will inform the patient about the study, provide the information sheet, and obtain informed consent for participation in the study and data processing. Subsequently, the questionnaire will be used to interview the patients, collect their responses, and assign them to the corresponding level of palliative care (PC) according to the score obtained. The assignment to the level of PC intensity made by Pulmonologist A will not in any way modify the patient's allocation to the level of PC.

During the pulmonology visit, which takes place immediately after the questionnaire administration, Pulmonologist B will conduct the visit according to the standard procedures (collection of past medical history, recent history, occupational history, family history, evaluation of laboratory and instrumental tests, medical examination, measurement of viral parameters, potential prescription of antifibrotic medication, and oxygen therapy if respiratory failure is detected, etc.). At the end of the visit, Pulmonologist B will give their clinical judgment on the appropriate level of PC required for the patient, based on the visit and collected data.

On the same day, the patient will also have an appointment with the PC team (doctor and nurse), as per current protocols at APPI Fibrosi IRCCS AOUBO, during which information on the patient's symptoms, the impact of symptoms on daily life activities, quality of life (QoL), and the patient's support network will be gathered. At the end of the visit, the PC team will express their judgment on the referral of a patient to a specific level of PC, based on the visit and collected data.

As per clinical practice, Pulmonologist B can give their own opinion, but the final decision regarding the assignment is made by the PC team.

The questions administered through the questionnaire were formulated based on elements identified during the clinical practice of pulmonologists and the dedicated nurse of the APPI Fibrosi unit at the IRCCS. These elements are considered most likely to be associated with the need for a higher level of palliative care (PC), namely:

Use of oxygen therapy: This implies the presence of underlying organ failure (respiratory failure) and often constitutes an obstacle for patients leaving their homes, either due to induced depressive and/or anxious states or due to difficulties-especially among elderly patients-in using oxygen therapy devices. IPF is a disease often complicated by the development of chronic partial respiratory failure. Patients are thus at risk of chronic hypoxia and receive long-term home oxygen therapy prescriptions. Although there is no specific literature on adherence to chronic oxygen therapy in IPF patients, it can be assumed to be similar to that observed in patients with other chronic respiratory diseases. In a cohort of patients with chronic obstructive pulmonary disease (COPD), overall adherence to oxygen therapy was 60%, dropping further among those prescribed 24-hour therapy. An Italian study on COPD patients found that only 40% used portable oxygen devices to leave their homes, citing "shame" as the primary limiting factor. We believe that many IPF patients similarly restrict their outings for the same reason.

Progressive exertional dyspnea: This is a common symptom in IPF patients, impacting their quality of life (QoL) over months and years. As the disease progresses, worsening dyspnea makes even minimal physical activities difficult, affecting various aspects of life, including family relationships and social participation. Therefore, we have decided to assign a higher score to patients with greater dyspnea levels, as measured by the modified Medical Research Council (mMRC) scale. The mMRC scale is structured as follows:

mMRC 0: Dyspnea with strenuous exertion. mMRC 1: Dyspnea with moderate-to-intense exertion (e.g., brisk walking or running on level ground or slight incline).

mMRC 2: Dyspnea with moderate exertion (e.g., slower walking on level ground compared to peers or needing to stop during normal-paced walking).

mMRC 3: Dyspnea with light exertion (e.g., needing to stop to breathe after walking 100 meters or for a few minutes on level ground).

mMRC 4: Dyspnea at rest (e.g., experiencing dyspnea while dressing or undressing).

Difficulties in reaching the center (APPI Fibrosi) for logistical reasons or lack of caregiver support: Patients with such difficulties are more likely to refuse palliative care at the IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di S. Orsola, which puts them at risk of not receiving adequate support for managing symptoms associated with their underlying condition. On the other hand, home-based or community-based care presents an opportunity for those who would otherwise face challenges in accessing care.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* New diagnosis of Idiopathic Pulmonary Fibrosis (IPF) established through a Multidisciplinary Interstitial Disease Meeting.
* Obtaining written informed consent.

Exclusion Criteria:

* Patient's inability to understand and/or respond to the questions in the questionnaire as judged by the healthcare provider.
* Patient already receiving care from the Palliative Care Service.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of Idiopathic Pulmonary Fibrosis (IPF) established after discussion at the Multidisciplinary Interstitial Disease Meeting and referred to the APPI Fibrosi unit of the IRCCS for specialized care
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-09-19 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of concordance between the levels of palliative care obtained using a triage questionnaire and those derived from the clinical judgments of the dedicated pulmonologist and the dedicated palliative care physician | 18 months
  The primary objective will be measured by calculating Krippendorff's alpha coefficient of reliability among the classifications obtained with the questionnaire, the clinical judgment of the pulmonologist, and the clinical judgment of the palliative care physician

SECONDARY OUTCOMES:
Description of the degree of palliative care needs that patients with IPF present when referred to the reference pulmonology center | 18 months
  The secondary objective will be measured by calculating the percentage of patients assigned to each level of palliative care (PC) by the questionnaire, the pulmonologist, and the palliative care physician, as well as the number of patients who, at the time of formal IPF diagnosis, require a high level of palliative care according to the judgment of the pulmonologist and the palliative care team

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Nava, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliera-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided